CLINICAL TRIAL: NCT05807802
Title: Association Between FSTL1 and Postoperative Pulmonary Complications on Pediatric Within Living Donor Liver Transplantation:a Prospective Cohort Analysis
Brief Title: FSTL1 and PPCs on Pediatric Within LDLT:a Prospective Cohort Analysis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tianjin First Central Hospital (Other)
Responsible Party: Principal Investigator, Yingli Cao, Principal investigator, Tianjin First Central Hospital
Other Study IDs: FSTL1 on PPC after LDLT
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Acute Lung Injury/Acute Respiratory Distress Syndrome (ARDS); Pulmonary Complication; Liver Transplant; Complications
Keywords: follistatins-like protein 1; pulmonary complication; living donor liver transplantation
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample immediately after induction of anesthesia (T1), 10 minutes at anhepatic stage (T2), 30 minutes at new hepatic stage (T3) and immediately after abdominal closure (T4)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to identify the association between FSTL1 elevation and acute lung injury (ALI) after pediatric liver transplantation.The main questions it aims to answer what the risk factors are for ALI in children and to evaluate the predictive value for the development of ALI.Participants will be divided into non-ALI group and ALI group according to whether they had ALI in a week after liver transplantation.Researchers will compare the difference between the two groups and use multivariate logistic regression analysis to screen the risk factors of ALI, and receiver operating characteristic(ROC) curve was used to evaluate the predictive efficacy of risk factors.

DETAILED DESCRIPTION:
Postoperative pulmonary complications(PPC) are complicated diseases with high morbidity and mortality for pediatric after living donor liver transplant (LDLT), Acute lung injury(ALI) after LDLT is a common and complex pulmonary complication, it is leading causes of disability and death,both in the acute and long-term postoperative period, the identification of effective prediction model involved in ALI is urgent and highly demanded.In order to observe the effect of follistim like protein 1(FSTL1) on the incidence of ALI who underwent LDLT, and explore the related mechanism, the investigators aim to collect more than 400 infant patients underwent LDLT from May 2023 to December 2023 in our single-center prospective study. Basic clinical data of children were recorded, including age, gender, alanine aminotransferase (ALT), aspartate aminotransferase (AST), International Normalized ratio (INR), childhood end-stage liver disease score (PELD) and other indicators.The expression levels of serum FSTL1 were recorded immediately after induction of anesthesia (T1), 10 minutes at anhepatic stage (T2), 30 minutes at new hepatic stage (T3) and immediately after abdominal closure (T4). Murray score was used to determine whether ALI occurred one week after LDLT, and the children were divided into non-ALI group and ALI group. Postoperative mechanical ventilation time, ICU stay time, total length of hospital stay and mortality during hospitalization are recorded.

The primary outcome utilised a regression approach to adjust for potential confounders associated with ALI and FSTL1. Multivariate logistic regression analysis was used to screen the risk factors of ALI, and ROC curve was used to evaluate the predictive efficacy of risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Patient was diagnosed with biliary atresia
* American society of anesthesiologists physical status Ⅱ-Ⅲ

Exclusion Criteria:

* Secondary liver transplantation or other important organ injury before surgery
* Present with congenital airway or respiratory malformation
* Acute respiratory infection or respiratory insufficiency was present within 1 month before surgery

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children who needed elective parental liver transplantation due to biliary atresia
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
the incidence of acute lung injury | 1 week after living donor liver transplantation
  Murray score was scored from four aspects: chest X-ray, hypoxemia score, positive end-expiratory pressure and lung compliance. The total score was the sum of the scores of all parameters the sum of the number of parameters adopted. The higher the score, the more serious the injury was.

SECONDARY OUTCOMES:
the expression level of serum FSTL-1 | immediately after induction of anesthesia (T1), 10 minutes at anhepatic stage (T2), 30 minutes at new hepatic stage (T3) and immediately after abdominal closure (T4)]
  Real-time fluorescence quantitative polymerase chain reaction (RT-qPCR) was used to detect the expression of FSTL-1 in serum